CLINICAL TRIAL: NCT03624400
Title: Internet-delivered Cognitive Behaviour Therapy for Sleep Problems in Adolescents with Autism Spectrum Disorder
Brief Title: Internet-delivered Cognitive Behaviour Therapy for Sleep Problems in ASD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stockholm University (Other)
Responsible Party: Principal Investigator, Nora Choque Olsson, PhD, Principal investigator, Stockholm University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Sleep Good Autism
Record Dates: First submitted 2018-06-23; First posted 2018-08-10 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Autism Spectrum Disorder; Sleep Disturbance; Insomnia
Keywords: Autism spectrum disorder; Sleep; Cognitive-behavioral treatment; Internet delivered treatment
MeSH Terms: conditions — Autism Spectrum Disorder; Parasomnias; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Internet-based CBT-I (Experimental): N= 120 participants are offered Internet-based Cognitive behaviour therapy for insomnia (CBT-I)
  Interventions: Behavioral: Internet-based CBT-I
- Internet-based psychoeducation (Active Comparator): N= 120 participants are offered Internet-based psychoeducation about sleep problems in ASD.
  Interventions: Behavioral: Internet-based psychoeducation

INTERVENTIONS:
Behavioral: Internet-based CBT-I — The adapted Internet-based CBT-I for adolescents with ASD includes sleep hygiene, restriction of time in bed, stimulus control, cognitive therapy, and relaxation techniques. The treatment consists of 8 weekly modules and each module consists of several website pages that will be presented in a fixed order, with preprogrammed modules containing information, interactive questionnaires, descriptions of exercises and movies.
  Arms: Internet-based CBT-I
Behavioral: Internet-based psychoeducation — Internet-based psychoeducation contains information about ASD, sleep difficulties and aspects of sleep hygiene. The intervention takes place in 8 weeks modules.
  Arms: Internet-based psychoeducation

SUMMARY:
This trial investigates the behavioural effects of Internet-based Cognitive behaviour therapy for insomnia (CBT-I) in adolescents with autism spectrum disorder with sleep problems. This is a randomised controlled trial.

DETAILED DESCRIPTION:
Sleep problems are common in adolescents with autism spectrum disorder (ASD)1. Internet-based Cognitive behaviour therapy for insomnia (iCBT-I) is considered as an evidence-based treatment for insomnia 2. To date, no Internet-based CBT-I delivered treatment for sleep problems in adolescents with ASD has been undertaken. The objective of the study is to investigate the efficacy and effectiveness of the Internet-based CBT-I for sleep problems in adolescents with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents with a clinical ASD diagnosis based on the Diagnostic and Statistical Manual-fifth edition (DSM-5). Participants have been investigated with the Autism Diagnostic Observation Schedule (ADOS).
* Insomnia diagnosis or sleep problems according to DSM-5
* Intelligence quotient (IQ) > 70 according to Wechsler Intelligence Scale for Children - fourth edition
* Psychiatric comorbidities according to DSM-5: anxiety disorders or depression.

Exclusion Criteria:

* The presence of clinically assessed self-injury
* High risk of suicidal behaviour
* borderline personality disorder or any form of schizophrenia or related disorders;
* substance abuse as well as physical illness or condition that was largely influence sleep condition.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in sleep impairment by using The Insomnia Severity Index (ISI) | Baseline, post intervention (8 weeks), 3 months post intervention follow-up and 6 months post intervention follow-up
  The ISI is a seven-item measure that yields a quantitative index of sleep impairment and treatment outcome. Participants rate the following components on a 5-point Likert scale ranging from 0 (not at all) to 4 (extremely): (a) severity of sleep-onset, sleep-maintenance, and early morning awakening problems; (b) satisfaction with current sleep pattern; (c) interference with daily functioning; (d) noticeability of impairment attributed to the sleep problem; and (e) level of distress caused by the sleep problem. Total scores range from 0 to 28, with higher scores indicating greater perceived insomnia severity.

SECONDARY OUTCOMES:
Sleep diaries by using Actigraphy | Baseline, post intervention (8 weeks), 3 months post intervention follow-up and 6 months post intervention follow-up
  An actigraph is a small instrument worn on the wrist or ankle to measure body movement and nighttime sleep parameters.
Quality of sleep by using Athens Insomnia Scale (AIS) | Baseline, post intervention (8 weeks), 3 months post intervention follow-up and 6 months post intervention follow-up
  AIS is a self-administered questionnaire assessing the quality of sleep.
Everyday functioning by using Developmental disabilities modification of the Children's Global Assessment scale (DD-CGAS) | Baseline, post intervention (8 weeks), 3 months post intervention follow-up and 6 months post intervention follow-up
  The DD-CGAS is an instrument used by clinicians to rate patients' global everyday functioning.
Anxiety problems by using Spence Children's Anxiety Scale | Baseline, post intervention (8 weeks), 3 months post intervention follow-up and 6 months post intervention follow-up
  The SCAS is a 38-item parent report measure of children's anxiety.
Emotion regulation difficulties by using The brief version of Difficulties in Emotion Regulation Scale (DERS-16) | Baseline, post intervention (8 weeks), 3 months post intervention follow-up and 6 months post intervention follow-up
  The DERS-16 is a brief version of self-report measure of emotion regulation difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Nora Choque Olsson, PhD, Principal Investigator — Stockholm University
Locations (1):
- Nora Choque Olsson, Stockholm, Sverige, Sweden

REFERENCES:
- [Background] Owens J. Classification and epidemiology of childhood sleep disorders. Prim Care. 2008 Sep;35(3):533-46, vii. doi: 10.1016/j.pop.2008.06.003. PMID 18710669
- [Background] Bastien CH, Morin CM, Ouellet MC, Blais FC, Bouchard S. Cognitive-behavioral therapy for insomnia: comparison of individual therapy, group therapy, and telephone consultations. J Consult Clin Psychol. 2004 Aug;72(4):653-9. doi: 10.1037/0022-006X.72.4.653. PMID 15301650
- [Background] Georen L, Jansson-Frojmark M, Nordenstam L, Andersson G, Olsson NC. Internet-delivered Cognitive Behavioral Therapy for insomnia in youth with autism spectrum disorder: A pilot study. Internet Interv. 2022 May 23;29:100548. doi: 10.1016/j.invent.2022.100548. eCollection 2022 Sep. PMID 35651733